CLINICAL TRIAL: NCT05828186
Title: Calcification Remodeling Utilizing Shockwave LiThotripsy in Coronary Artery CaLcification (Guangxi Real-World Study)
Brief Title: CRUSTAL Study in China
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: IC-ISR001
Record Dates: First submitted 2023-04-01; First posted 2023-04-25 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease; Calcification
MeSH Terms: conditions — Coronary Artery Disease; Calcinosis | interventions — Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Shockwave Coronary Intravascular Lithotripsy (IVL) catheter — Patients with coronary artery calcification who are planned to undergo PCI and are deemed in need of Shockwave IVL catheter treatment by their physicians.

SUMMARY:
This is a prospective, multicenter, single-arm registry study, aimed to evaluate the clinical outcomes of using Shockwave IVL catheter in the treatment of coronary artery calcification in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Patients with coronary artery calcification who are planned to undergo PCI and are deemed in need of Shockwave IVL catheter treatment by their physicians.
* The subject or their legal representative agrees to sign the informed consent form.

Exclusion Criteria:

* The physician evaluates that the subject's expected lifespan is <1 year.
* The subject did not receive IVL treatment in the index procedure.
* The subject is pregnant or lactating.
* The subject is currently participating in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with coronary artery calcification who are planned to undergo percutaneous coronary intervention (PCI) and are deemed suitable to receive Shockwave IVL catheter treatment by their physicians.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedure success | in 48 hours post-procedure or prior to discharge, whichever comes first
  Procedure success defined as successful stent implantation, residual stenosis degree <30% (core laboratory), and no major adverse cardiac events (MACE) occurring during hospitalization
Freedom from major adverse cardiac events (MACE) within 30 days of the index procedure | 30 days post index procedure
  MACE is defined as:
  Cardiac death; or Myocardial Infarction (MI): Follow the Fourth Universal Definition of Myocardial Infarction ; or Target Vessel Revascularization (TVR) defined as revascularization at the target vessel (inclusive of the target lesion) after the completion of the index procedure; or Target lesion thrombosis.

SECONDARY OUTCOMES:
Vascular complications in the proudure | Immediately post index procedure
  Vascular complications is defined as:
  Perforation or Severe dissection or Acute occlusion or Consistent No-reflow/ slow flow
Incidence of target lesion revascularization | 30 days post index procedure
Incidence of target lesion revascularization | 6 months post index procedure
30 days post index procedure | 9 months post index procedure
Incidence of target lesion revascularization | 12 months post index procedure

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - liuzhou People's Hospital, Liuchow, Guangxi
  - Yulin First People's Hospital, Yulin, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanjing, Guanxi
  - Guilin People's Hospital, Guilin
  - Guiping People's Hospital, Guiping
  - Liuzhou labors' Hospital, Liuchow

IPD SHARING:
Plan to Share IPD: Undecided